CLINICAL TRIAL: NCT03482921
Title: Body Parameters as an Independent Predictor of Acute Pancreatitis: A Propensity Score-matched Case-control Study
Brief Title: Body Parameters as an Independent Predictor of Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ningbo4
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to assess the predictive significance of visceral adipose tissue (VAT) and visceral adipose tissue /skeletal muscle tissue ratio (VAT/SMT ratio) for the prognosis in acute pancreatitis (AP) patients.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a sudden inflammation of the pancreas. However, one-fifth of patients may develop severe complications with a mortality between 10%-20% It remains a difficulty to find an effective method for prediction of severity of AP at early stage.

It is well-established that obesity (defined as body mass index[BMI]>30kg/m2 by the World Health Organization) is a risk factor for AP and increases the incidence of systemic complication, motality. There are a lot of parameters related to saropenic obesity, including areas of visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT), skeletal muscle tissue (SMT), and VAT/SMT ratio. it is unclear which parameter is the best predictor of severe AP. Thus, this study is aimed to investigate the association between these parameters and AP severity and find the best predictor of AP.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with AP
2. age >18 years

Exclusion Criteria:

1. age<18years
2. missing data in the electronic medical record
3. history of AP

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosis criteria for AP was defined as the presence of at least 2 of the 3 following factors: (1) abdominal pain characteristic of AP; (2) serum amylase and/or lipase levels≥3 times the upper limit of the normal level, and (3) characteristic findings of AP on a CT scanning.
Sampling Method: Non-Probability Sample
Enrollment: 1662 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Comparisons of variables according to AP severity | the physical examination data in the year of 2017
  Comparisons of variables according to AP severity by one-way analysis of variance (ANOVA) and Likelihood Ratio
Relationships between VAT and severity outcomes Relationships between VAT and severity outcomes Relationships between VAT and severity outcomes Relationships between body parameters and severity outcomes | the physical examination data in the year of 2017
  Relationships between VAT and severity outcomes by Likelihood Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xu, Dr, Principal Investigator — Department of gastroenterology, Ningbo No.1 Hospital, Ningbo, China
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Xie J, Xu L, Pan Y, Li P, Liu Y, Pan Y, Xu L. Impact of visceral adiposity on severity of acute pancreatitis: a propensity score-matched analysis. BMC Gastroenterol. 2019 Jun 13;19(1):87. doi: 10.1186/s12876-019-1015-z. PMID 31195984